CLINICAL TRIAL: NCT06259448
Title: Feasibility of Optimizing Organized Cervical Cancer Screening by Urine Self-sampling
Acronym: PAPPEES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/63
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; screening; urine self-sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- urine self-sampling (Experimental): urine self-sampling
  Interventions: Other: urine self-sampling

INTERVENTIONS:
Other: urine self-sampling — urine self-sampling

SUMMARY:
This project addresses the issue of promoting organized cervical cancer screening (CCS) from the perspective of the use of urine self-sampling (USS). Via a prospective and monocentric study, the present study aims to evaluate the acceptability of women to collect a urine self-sample and to respond to a questionnaire on their feelings about this screening method.

DETAILED DESCRIPTION:
In France, individual cervical cancer screening (CCS) has reduced the annual frequency of cervical cancer (CC), both in terms of incidence (2920 cases) and mortality (1117 deaths) : 2.5% reduction in CC incidence was observed per year between 1980 and 2012. More than 6 millions CCS are performed each year leading to the diagnosis of approximately 170,000 cytological abnormalities, including about 15,000 high-grade intraepithelial lesions, precursors of cancer. Since 2019, CCS is now recommended in France with cytology-based screening before 30 and high risk Human Papillomavirus (HPV) testing from 30 to 65 years-old (screening interval of 5 years after a negative test).

Since only 50 to 60% of the target population is currently screened, the French High Authority for Health (HAS) has recently recommended the implementation of an organized screening program (OSP) to increase screening-participation and to reduce inequalities in access to screening. This OSP includes sending an invitation to under screened women for a consultation and a clinician taken cervical sample. However, the response rate to the OSP of cancers to a first letter of invitation is generally low, less than 20% (for example, the rate of participation in colon cancer screening in the french department of Gironde is 18.8% in 2020 (data from French Regional Coordination Center for Cancer Screening). This trend is particularly true in rural areas with low medical density: northern and southern areas of Gironde are concerned with 2/3 of under-screened women for CCS. Reducing social and territorial inequalities in participation in organized CCS and optimizing the screening process for the least participating women remain a challenge.

Self-sampling kits, with the possibility to be sent to the women, seem to be a promising alternative to overcome the low participation in these areas.

Vaginal self-sampling has already been shown to increase participation. More recent studies have focused on urine self-sampling for the detection of cervical precancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 31 to 49
* Coming to the Bordeaux University Hospital for a gynecological consultation in order to have a cervical swab (PCC) for screening or follow-up.
* Patient affiliated to or benefiting from a social security system
* Non-objection to study participation

Exclusion Criteria:

* Patient unable to speak French and/or illiterate
* Patient under legal protection

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Urine self-sampling acceptability | Baseline
  Acceptability rate of self-testing obtained via questionnaire: The questionnaire survey methodology enables both quantitative and qualitative qualitative analysis of practices, opinions and behaviors according to and behaviors according to respondent characteristics (age, gender, level of education...). level, etc.). Content analysis of responses to open-ended questions consists in creating categories and classifying the different discourses in these categories categories in order to identify the main themes. The level of satisfaction will be assessed by classifying the emerging categories according to positive perceptions and obstacles.

SECONDARY OUTCOMES:
Cervical swab result | Baseline
  positive/negative
Urine test result | Baseline
  positive/negative

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No